CLINICAL TRIAL: NCT00697905
Title: An Open Labeled, Multicentre, Randomized Phase II Trial of Combination Gemcitabine and Carboplatin Chemotherapy in Patients With Metastatic or Recurrent Nasopharyngeal Carcinoma
Brief Title: Combination of Gemcitabine and Carboplatin in Metastatic or Recurrent Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Dr. Christina Ng Van Tze, University of Malaya Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT 06-01
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2010-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; Gemcitabine-Carboplatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Carboplatin; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Gemcitabine; Drug: Carboplatin
- B (Active Comparator)
  Interventions: Drug: Cisplatin; Drug: 5-fluorouracil (5-FU)

INTERVENTIONS:
Drug: Gemcitabine — Intravenous administration on days 1, 8 of a 21-day cycle
  Arms: A
Drug: Carboplatin — Intravenous following Gemcitabine infusion on day 1
  Arms: A
Drug: Cisplatin — Intravenous on day 1 prior to 5-FU infusion on days 2 to 5 of a 28-day cycle
  Arms: B
Drug: 5-fluorouracil (5-FU) — Intravenous infusion on day 2 to day 5
  Arms: B

SUMMARY:
The aim of the study is to assess if gemcitabine in combination with carboplatin as 1st line chemotherapy in patients with metastatic or recurrent nasopharyngeal carcinoma has reasonable efficacy and a favourable toxicity profile that warrants further comparative study. A parallel group of randomly selected patients of equal number to the carboplatin and gemcitabine combination arm will be treated with the cisplatin and 5-FU combination chemotherapy (active control arm).

The hypothesis is that this combination of chemotherapy is at least as active and less toxic than the reference regimen of cisplatin in combination with 5-fluorouracil (5-FU).

DETAILED DESCRIPTION:
52 patients with metastatic or recurrent nasopharyngeal carcinoma who meet inclusion/exclusion criteria will be enrolled into the trial. After initial screening, patients will attend clinic for baseline examination. Subjects will then be randomly allocated to carboplatin and gemcitabine or cisplatin and 5-FU combinations in a ratio of 1:1. Study visits will occur depending on which arm the patient is on.

An economic evaluation of the costs and benefits of gemcitabine-carboplatin will be implemented within this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from patient or parents/guardian.
2. Subject age greater than or equal to 18 years
3. Histologically proven recurrent or metastatic undifferentiated or squamous nasopharyngeal carcinoma, not amenable to local therapy.
4. Measurable disease in distant sites and/or loco-regional sites defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded as >=10mm with CT scan or MRI. Tumour lesions that are situated in a previously irradiated field are measurable only if the tissue planes are preserved on CT or MRI).
5. Prior concurrent chemotherapy and radiation therapy is permitted.
6. Primary chemo-radiotherapy must be completed at least 6 months prior to study entry.
7. Life expectancy over 3 months.
8. ECOG performance status less than or equal to 2.
9. Patients must have normal organ and marrow function as follows:

   * White blood cell count : >= 3.0 x 10^9/L
   * Absolute neutrophil count : >= 1.5 x 10^9/L
   * Platelets : >= 100 x 10^9/L
   * Total bilirubin : within normal limits
   * AST/ALT/ALP : <= 2.5 x upper limit of normal
   * Creatinine clearance or estimated GFR : >=50 mls/min.

Exclusion Criteria:

Patients with any of the following are not eligible for enrollment into the study:

1. Pregnant women are excluded from this study because gemcitabine has potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with gemcitabine, breastfeeding should be discontinued if the mother is treated with gemcitabine. These potential risks may also apply to other agents used in this study.
2. Women of child-bearing potential and men without an adequate contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
3. Prior use of gemcitabine
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine or carboplatin.
5. Prior lines of chemotherapy for metastatic NPC
6. Prior radiotherapy to the indicator lesion(s) to be measured in the study.
7. Patients receiving any other investigational agents
8. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
9. Patients with bone-only metastases.
10. Clinically significant cardiac disease (e.g. congestive cardiac failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
11. Severe sensorineural hearing loss affecting normal daily activities or requiring the use of hearing aids.
12. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
13. Patients with immune deficiency. They are at increased risk of lethal infections when treated with marrow-suppressive therapy.
14. HIV-positive patients receiving combination antiretroviral therapy. There is a possible pharmacokinetic interaction between antiretroviral and gemcitabine or other agents administered during the study. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is response to therapy. Response will be evaluated using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. | 12 months

SECONDARY OUTCOMES:
Progression free survival defined as the duration of time from start of treatment to time of disease progression or death, whichever occurs first. | 12 months
Duration of response defined as the interval between the first documented response (CR or PR) and the first documented sign of disease progression or death, whichever occurs first. | 12 months
Safety and tolerability assessments will consist of 1.Monitoring and recording all AE and SAE, 2.Regular monitoring of hematology, blood chemistry and urinary laboratory parameters, 3.Regular performance of physical examinations, including vital signs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christina Ng, Principal Investigator — University of Malaya
Locations (11):
- Malaysia (11):
  - Loh Guan Lye Specialist Centre, George Town
  - Penang General Hospital, George Town
  - Ipoh Specialist Centre, Ipoh
  - Johor Specialist Centre, Johor Bahru
  - NCI Cancer Hospital, Kampung Baharu Nilai
  - Likas Hospital, Kampung Likas
  - Sabah Medical Centre, Kota Kinabalu
  - Tung Shin Hospital, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Universiti Sains Malaysia, Kubang Kerian
  - Normah Medical Specialist Centre, Kuching

REFERENCES:
- See also: Related Info — http://www.crc.gov.my